CLINICAL TRIAL: NCT05723718
Title: MalnutritiOn Assessment With biOelectrical impedaNce Analysis in gastRic Cancer patIentS Undergoing Multimodal trEatment - MOONRISE Study
Brief Title: MalnutritiOn Assessment With biOelectrical impedaNce Analysis in gastRic Cancer patIentS Undergoing Multimodal trEatment
Acronym: MOONRISE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Lublin (Other)
Collaborators: Erasmus Medical Center (Other); Ohio State University (Other); Poznan University of Medical Sciences (Other); Jagiellonian University (Other)
Responsible Party: Sponsor
Other Study IDs: MOONRISE_2023
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Malnutrition; Cachexia
Keywords: gastric cancer; bioelectrical impedance analysis; body composition; nutritional status; malnutrition; cachexia; multimodal treatment; tumor regression grade
MeSH Terms: conditions — Stomach Neoplasms; Malnutrition; Cachexia | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Survey — Evaluation of the nutritional status and body composition on tumor regression grade in gastric cancer patients scheduled for multimodal treatment. Nutritional status assessment will include: selected clinical variables evaluation (weight, BMI, nutritional status scales), bioelectrical impedance analysis and selected laboratory parameter assessment. After inclusion in the study, each patient will have four consecutive nutritional status assessments: (1) one day prior staging laparoscopy or during qualification to neoadjuvant chemotherapy, (2) one day before the gastrectomy, (3) one month after the gastrectomy, (4) after the last cycle of adjuvant chemotherapy.
  Other Names: Nutritional Status and Body Composition Assessment

SUMMARY:
The aim of this single-arm prospective, multicenter, cross-sectional study is to evaluate the nutritional status and body composition on tumor regression grade with bioelectrical impedance analysis in gastric cancer patients undergoing multimodal treatment. Results of this study will reveal whether nutritional status and body composition assessment based on bioelectrical impedance analysis will become a validated and objective tool to support clinical decisions in gastric cancer patients undergoing multimodal treatment.

DETAILED DESCRIPTION:
Up to 20% of gastric cancer patients experience unintentional loss of their pretreatment body weight. Malnutrition contributes to increased morbidity, higher risk of perioperative complications and systemic toxicity. A standardized approach to evaluate the nutritional status of gastric cancer patients is yet to be established. Bioelectrical impedance analysis is a non-invasive technique estimating changes in body composition over time.

125 patients with locally advanced gastric adenocarcinoma scheduled for multimodal treatment will be included in the study. Four consecutive nutritional status assessments will be performed throughout the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed gastric adenocarcinoma (or undifferentiated carcinoma)
3. Stage II - III disease (cT2 cN+ and cT3-T4 cN+/-) based on the 8th edition of TNM classification
4. Qualification for multimodal treatment by the decision of the multidisciplinary tumor board

Exclusion Criteria:

1. Early gastric cancer (cT1N0-3M0) scheduled for endoscopic treatment by multidisciplinary team
2. Gastric stump carcinoma
3. Distant metastasis
4. Upfront surgery
5. Other malignancies
6. Contraindications to bioelectrical impedance analysis (e.g., implanted cardiac devices, metal implants or pregnancy)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a western population of patients with histologically confirmed, potentially curative esophageal gastro junction and gastric adenocarcinoma scheduled for multimodal treatment.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Regression Grade | Up to 2-4 weeks after the surgery
  determined using the Becker criteria (1- complete response, 2 - good response, 3 - partial response, 4 - no response)

SECONDARY OUTCOMES:
Neoadjuvant Chemotherapy Toxicity | From date of inclusion up to 1-3 months after the date of the first neoadjuvant chemotherapy cycle
  evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) criteria (version 5.0)
Postoperative Complications | From date of surgery, assessed up to 90 days
  Assessed by the Comprehensive Complication Index (CCI). Min-Max values (0-100), higher scores mean a worse outcome
Overall Survival | From from the date of surgery to the date of patient death or the date of the last follow-up - up to 10 years
  Overall survival analysis will determine whether bioelectrical impedance analysis is a prognostic factor in advanced gastric cancer patients
Quality of Life score | From date of inclusion through study completion - an average of 3 years
  Assessment based on The European Organization for Research and Treatment of Cancer quality of life, gastric-cancer specific questionnaire(EORTC QLQ - STO22). Min-Max value (1-7); higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zuzanna Pelc, PhD, Principal Investigator — Medical University of Lublin
Locations (1):
- Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pelc Z, Sedlak K, Mlak R, Chawrylak K, Mielniczek K, Lesniewska M, Skorzewska M, Kwietniewska M, Pasnik I, Geca K, van der Sluis P, Banasiewicz T, Pedziwiatr M, Polkowski WP, Pawlik TM, Malecka-Massalska T, Rawicz-Pruszynski K. MalnutritiOn assessment with biOelectrical impedaNce analysis in gastRic cancer patIentS undergoing multimodaltrEatment (MOONRISE)-Study protocol for a single-arm multicenter cross-sectional longitudinal study. PLoS One. 2024 Feb 6;19(2):e0297583. doi: 10.1371/journal.pone.0297583. eCollection 2024. PMID 38319910